CLINICAL TRIAL: NCT01076296
Title: A Post-Marketing Study for On Label Evaluation of the GE Vscan Ultrasound Imaging System
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: OHSU_Vscan_02
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Left Ventricular Dysfunction; Right Ventricular Dysfunction; Pulmonary Hypertension; Heart Valve Diseases
MeSH Terms: conditions — Ventricular Dysfunction, Left; Ventricular Dysfunction, Right; Hypertension, Pulmonary; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to collect data and learn more about the Vscan Ultrasound Imaging System. It is an "observational" study with no additional procedures or intervention prescribed other than using the Vscan along with a routine medical physical exam.

DETAILED DESCRIPTION:
The study requires 2 visits to OHSU.

At the first visit a cardiac physical exam will be done by a cardiologist.

At a second visit, a different cardiologist will perform an ultrasound scan (as part of your standard of care) using a Vscan Ultrasound System. The first and the second visit may be done on the same day depending upon your schedule and if it's convenient for you to stay. The total exam time for both the visits, including standard exam and the study device exam will be about 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* provided signed and dated informed consent and is willing to provide GE Healthcare with demographic data, cardiac medical history, information collected as part of the study
* New patients who have an echocardiogram less than 6 months and patients who will be undergoing an echocardiogram as part of their routine clinical care

Exclusion Criteria:

* Pregnant
* less than 18 years of age.
* unwilling to provide informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-patient and outpatient population of OHSU Division of Cardiovascular Medicine
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Kaul, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Abnormal Left Ventricle Function: Subjects assessed for LV function with both VScan and a clinical examination noting an abnormality.
- Normal Left Ventricle Function: Subjects assessed for LV function with both VScan and a clinical examination noting no abnormality.
- Abnormal Right Ventricle Function: Subjects assessed for RV function with both VScan and a clinical examination noting an abnormality.
- Normal Right Ventricle Function: Subjects assessed for RV function with both VScan and a clinical examination noting no abnormality.
- Pulmonary Hypertension: Subjects assessed for Pulmonary Hypertension with both VScan and a clinical examination noting the presence of pulmonary hypertension.
- No Pulmonary Hypertension: Subjects assessed for Pulmonary Hypertension with both VScan and a clinical examination noting no presence of pulmonary hypertension.
- Heart Valve Disease: Subjects assessed for HVD with both VScan and a clinical examination noting the presence of HVD.
- No Heart Valve Disease: Subjects assessed for HVD with both VScan and a clinical examination noting no presence of HVD.
Period: Overall Study
Arm/Group | Abnormal Left Ventricle Function | Normal Left Ventricle Function | Abnormal Right Ventricle Function | Normal Right Ventricle Function | Pulmonary Hypertension | No Pulmonary Hypertension | Heart Valve Disease | No Heart Valve Disease
Started | 54 | 196 | 51 | 199 | 59 | 191 | 51 | 199
Completed | 54 | 196 | 51 | 199 | 59 | 191 | 51 | 199
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total for All Groups Assessed: Subjects assessed for LV function using both VScan and a clinical examination.
Arm/Group | Total for All Groups Assessed
Number analyzed (Participants) | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 656
  Male | 344

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Correct Diagnosis
Description: A comparison of the percentages of correct diagnosis by VSCAN and clinical exam using a McNemar test for matched pairs with ECHO used as the gold standard.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of correct diagnosis
Groups:
- Pulmonary Hypertension: Subjects assessed for Pulmonary Hypertension function with both VScan and a clinical examination noting the presence of pulmonary hypertension.
- No Pulmonary Hypertension: Subjects assessed for Pulmonary Hypertension function with both VScan and a clinical examination noting the no presence of pulmonary hypertension.
- Heart Valve Disease: Subjects assessed for Heart Valve Disease function with both VScan and a clinical examination noting the presence of HVD.
- No Heart Valve Disease: Subjects assessed for Heart Valve Disease function with both VScan and a clinical examination noting no presence of HVD.
Arm/Group | Abnormal Left Ventricle Function | Normal Left Ventricle Function | Abnormal Right Ventricle Function | Normal Right Ventricle Function | Pulmonary Hypertension | No Pulmonary Hypertension | Heart Valve Disease | No Heart Valve Disease
Number analyzed (Participants) | 54 | 196 | 51 | 199 | 59 | 191 | 51 | 199
percentage of correct diagnosis | 61 [45 to 77] | 31 [23 to 39] | 47 [26 to 67] | 6 [1 to 12] | 10 [8 to 29] | 3 [3 to 9] | 39 [19 to 59] | 4 [2 to 9]

ADVERSE EVENTS:
Arm/Group | Abnormal Left Ventricle Function | Normal Left Ventricle Function | Abnormal Right Ventricle Function | Normal Right Ventricle Function | Pulmonary Hypertension | No Pulmonary Hypertension | Heart Valve Disease | No Heart Valve Disease
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/196 | 0/51 | 0/199 | 0/59 | 0/191 | 0/51 | 0/199
Other Adverse Events (participants affected / at risk) | 0/54 | 0/196 | 0/51 | 0/199 | 0/59 | 0/191 | 0/51 | 0/199

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less